CLINICAL TRIAL: NCT04338594
Title: Impact of the Profession on Parenthood
Acronym: MEDparenting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2020 MEDparenting
Record Dates: First submitted 2020-04-04; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-03

CONDITIONS: Parenthood Status
Keywords: Parenthood; Work; child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Professional constraints can have major causes on personal and couple life. In particular, some professions with major professional constraints that can be particularly impacted, such as doctors and healthcare workers.

The main objective was to demonstrate the impact of work on the desire and the fact to have children

DETAILED DESCRIPTION:
This is an observational study by questionnaire via an internet link. The self-questionnaire will assess parenthood, socio-demographic parameters, and the perception of the profession.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers
* Workers or retirees

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Workers or retirees
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
parenthood | Day 1
  The desire to have a child and the parenting management will be assessed by questionnaires

SECONDARY OUTCOMES:
Sociodemographic characteristics | Day 1
  Age, gender, qualification, personal work status, ethnicity, life and occupational events will be assessed by questionnaires
occupation perception | Day 1
  the perception about occupation will be assessed by questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, Clermont-Ferrand, Clermont-Ferrand, France